CLINICAL TRIAL: NCT05778097
Title: Adjuvant Androgen Deprivation Therapy Combined With Apalutamide for Prostate Cancer Patients Post Radical-prostatectomy With High-risk of Reoccurrence: a Prospective, Single-arm, Multicenter Trial (ARES Study)
Brief Title: Adjutant Apalutamide Plus ADT in Post-RP Patients With High Risk of Recurrence (ARES Study)
Acronym: ARES
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Principal Investigator, Hongqian Guo, Chief physician of Department of Urology, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-115
Record Dates: First submitted 2023-03-04; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer; Biochemical Recurrence; High Risk
Keywords: prostate cancer biochemical recurrence; apalutamide; adjuvant treatment; post-radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apalutamide+ADT (Experimental): Apalutamide (240 mg once daily) in combination with ADT for 12 cycles (28 days of each cycle)
  Interventions: Drug: Apalutamide 60mg Tab; Drug: Androgen deprivation therapy(ADT)

INTERVENTIONS:
Drug: Apalutamide 60mg Tab — Apalutamide 60Mg Tab (4 x 60 mg) once daily on days 1-28 of a 28-day cycle
Drug: Androgen deprivation therapy(ADT) — The choice of ADT will be at discretion of the Investigator. Dosing (dose and frequency of administration) will be consistent with the prescribing information.

SUMMARY:
ARES is a multicenter, single-arm, phase 2 trial to evaluate the efficacy and safety of ADT in combination with apalutamide as an adjuvant regimen for patients with high risk of recurrence after radical prostatectomy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Prostate cancer diagnosed histologically or cytologically in males ≥18 years and ≤75 years of age;
2. Localized prostate cancer (assessed by conventional imaging tools such as CT and bone scan) within 12 weeks after radical prostatectomy;
3. PSA < 0.1 ng/ml within 8 weeks after surgery;
4. Postoperative CAPRA-S score ≥ 6, suggesting a higher risk of recurrence;
5. ECOG score at 0-1 according to the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale;
6. Adequate organ functions:

   Hematology (within 14 days before treatment: no blood transfusion, no use of granulocyte colony-stimulating factor, no use of other drugs for correction)：
   1. Neutrophil count (NE) ≥1.5×109/L;
   2. Hemoglobin (HGB) ≥ 90 g/L;
   3. Platelet count (PLT) ≥100×109/L; Coagulation function (no blood product transfusion within 14 days before treatment): international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5× upper limit of normal (ULN); Blood biochemistry (liver and kidney function)：

   <!-- -->

   1. Creatinine clearance ≥ 30 mL/min;
   2. Total bilirubin (TBIL) ≤ 1.5× ULN;
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN;
7. Ability to provide written informed consent form (ICF) and ability to understand and agree to adhere to study requirements and schedule of assessments;
8. Patients of childbearing potential must be willing to use highly effective contraception during the study and for 12 weeks after the last dose of treatment.

Key Exclusion Criteria:

1. Patients with neuroendocrine, small cell, or sarcomatoid features in prostate histopathology;
2. Pelvic lymph node metastasis (cN1) or distant metastasis (cM1) indicated preoperatively by traditional imaging procedures such as CT or bone scan;
3. Prior treatment by androgen deprivation therapy (including medication or surgical castration), focal therapy for prostate cancer, or radiotherapy and chemotherapy for prostate cancer;
4. Prior treatment with second-generation antiandrogen (e.g., abiraterone, apalutamide, enzalutamide, darolutamide, etc.);
5. Any major surgery (other than radical resection) requiring general anesthesia within 28 days prior to the first dose of the study;
6. Other malignancies present or occurred in the past 2 years, except cured non-melanoma skin cancers and superficial bladder tumors (Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating of basement membrane);
7. Arterial/venous thrombotic events (such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism) or anticoagulant therapy with warfarin or heparin within 6 months before the study;
8. Corrected QT interval (QTc) of heart rate > 500 ms; patients with QTc prolonged but < 500 ms should be assessed by a cardiologist for eligibility;
9. Severe cardiovascular diseases: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia; Classes III-IV cardiac insufficiency according to the New York Heart Association (NYHA) Classification, or left ventricular ejection fraction (LVEF) < 50% indicated in cardiac Doppler ultrasound;
10. Allergy to any study drug or excipients;
11. Active viral hepatitis requiring treatment as determined by the Investigators:

    1. Chronic hepatitis B, with hepatitis B virus (HBV) deoxyribonucleic acid (DNA) ≥ 500 IU/mL (2500 copies/mL) (HBV DNA testing only for patients with positive test for Hepatitis B surface antigen or core antibody);
    2. Positive for Hepatitis C virus (HCV) ribonucleic acid (RNA) test (HCV RNA test only for patients with positive HCV antibodies);
12. Any present active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism), or known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation, or long-term heavy use of hormones or other immunomodulators, or other conditions assessed by the Investigator as having an impact on study treatment;
13. Active infection;
14. History of interstitial lung disease or uncontrolled systemic disease, including diabetes, hypertension, acute lung disease, etc.;
15. Known to have human immunodeficiency virus (HIV) infection;
16. History of epilepsy or conditions that may induce epilepsy
17. The presence of an underlying medical condition alcohol/drug abuse or dependence that is detrimental to the administration of the study drugs, or that may affect the interpretation of the results, or that places the patient at high risk of developing treatment complications;
18. Men who have sexual activity with women of childbearing potential, unless they:

    Agree to use condom or spermicidal foam/gel/diaphragm/cream/suppository Agree not to donate sperm during the study and for at least 3 months after receiving the last dose of study drug No birth plan during the study or within 3 months after the last dose of study drug
19. Concurrent participation in another therapeutic clinical study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Two-year biochemical progression-free survival | 24 months
  It is defined as the proportion of patients without biochemical progression or death 2 year after initiation with Apalutamide plus ADT.
  Biochemical progression is defined as an increase of more than 0.5 ng/mL from PSA nadir after treatment (confirmed rise on at least two separate occasions) or any evidence of clinical relapse/metastasis or the initiation of any anti-prostate cancer therapy or death due to any cause.

SECONDARY OUTCOMES:
Event-free survival rate | from initiation with apalutamide up to 36 months
  It is defined as the proportion of patients without biochemical recurrence or any evidence of clinical relapse/metastasis or initiation of any other anti-prostate cancer therapy or death due to any cause.
Biochemical progression-free survival | 60 months
  It is defined as the time from the initiation of treatment to the first occurrence of biochemical recurrence, and the definition of biochemical progression is the same as that of the primary observation endpoint;
Metastasis-free survival (MFS) | 60 months
  It is defined as the time from the start of treatment to the first occurrence of distant metastasis or death, whichever occurs first; distant metastasis can be diagnosed by imaging results or pathology by Blinded Independent Central Review (BICR);
Quality of life (QoL) assessed by FACT-P scale | 24 months
  The FACT-P scale (39 items) includes a Functional Assessment of Cancer Therapy - General (FACT-G, which consists of 4 subscales measuring physical, functional, social/family, and emotional well-being) and a specific subscale for prostate cancer. The total score is calculated by summing the scores of FACT-G and the prostate cancer subscales, ranging from 0 to 156, with higher scores indicating better functional status
Two-year testosterone recovery rate | 24 months
  It is defined as the proportion of patients with testosterone recovery 2 year after initiation of apalutamide plus ADT. Testosterone recovery is defined as testosterone level >50 ng/dL.
Time to testosterone recovery | From initiation of apalutamide plus ADT up to 36 months
  Testosterone recovery is defined as testosterone level >50 ng/dL
Number of Adverse Events Number of Adverse Events Number of Adverse Events Adverse events (AEs) | From initiation of apalutamide plus ADT to 30 days after last dose of apalutamide
  All adverse events (AEs) are assessed and graded according to NCI-CTCAE v5.0. Safety will be assessed and documented after the initiation of study drug, regardless of relationship to the study drug, until 30 days after the last study treatment or the initiation of new antineoplastic therapy, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nanjing Tumor Hospital, Nantong, Jiangsu

IPD SHARING:
Plan to Share IPD: No